CLINICAL TRIAL: NCT05646914
Title: Effect of Plyometric and Complex Training on Physical Performance in Male Cricket Players: a Randomized Controlled Trial
Brief Title: Plyometric and Complex Training in Male Cricket Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16.11.2015
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Physical Functional Performance
Keywords: Muscle strength; Fitness; Athletes; Exercise; Power
MeSH Terms: conditions — Motor Activity | interventions — Plyometric Exercise

STUDY DESIGN:
Intervention Model Description: A randomized control study with a pretest-posttest design.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor was kept blinded to allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Complex training group (Experimental): Plyometric exercises along with resistance exercises were performed.
  Interventions: Other: Complex training exercises
- Plyometric training group (Active Comparator): Plyometric exercises were performed.
  Interventions: Other: Plyometric training exercises
- Control group (No Intervention): Routine training was performed.

INTERVENTIONS:
Other: Complex training exercises — Squats and drop jumps, Barbell step-ups and hops, Bench press and plyometric press-up, Barbell lunge and box jumps were performed.
  Arms: Complex training group
Other: Plyometric training exercises — Drop Jumps, Hops, Plyometric press-up, Box Jumps were performed.
  Arms: Plyometric training group

SUMMARY:
The complex training starts with a high load of resistance training that is succeeded by plyometric training. This combination aims at improving the efficacy of the plyometric training stimulus, thus increasing the neuromuscular response, explosive strength, and power. This response might further be improved by making appropriate variations in the dosage parameters of complex training. Previously available literature reports conflicting evidence, with some studies supporting the effectiveness of complex training for improving power output in sports, whereas others contradict this rationale. There is a paucity of research evidence that directly compares the efficacy of plyometric and complex training for the outcomes of physical performance in cricket players.

ELIGIBILITY:
Inclusion Criteria:

* University-level cricket players
* Age of 18 to 26 years
* Playing competitively at least once a month
* Involved in resistance training for at least six months
* Working knowledge of the english language

Exclusion Criteria:

* A history of severe neurological deficit, injury or concussion in the past six months,
* Operative treatment for lower or upper limb in the past six months,
* Current musculoskeletal pain (any level of chronicity)

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-05-23 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Core Muscle Strength | 4 weeks.
  Athletes assumed a pike position with the elbows under the shoulders, the forearms shoulder-width apart on the floor, toes on the floor, buttocks in a neutral position, and the body in a straight line.
Multistage Fitness | 4 weeks.
  For this test, the subject had to run between two lines marked 66 feet apart (20 meters). Pre-recorded beeps were played, and the subjects had to increase their speed with each beep, thereby determining their aerobic fitness based on the number of laps completed.
Push-Up | 4 weeks.
  The subjects performed the push-up with their hands and toes touching the floor. In the eccentric phase, the subjects moved down until they were at a 5 cm distance from the floor. The total number of push-ups completed in proper form was counted.
Lateral Cone Jump | 4 weeks.
  Two cones were kept with a crossbar or tape fastened across them with the subject standing on one side. The subjects were made to jump to cross the bar and land on the opposite side. The time was started as soon as the subject's foot left the ground, and the total number of lateral jumps performed in 30 seconds was counted.
Stationary Vertical Jump | 4 weeks.
  A tape measure was attached to the wall, with the subject standing adjacent to it. They were supposed to touch the highest point on the wall with their inked middle fingertip. This point was taken as the standing height of the subject. Then, the subject performed a vertical jump with the assistance of both arms and legs to reach the maximum possible height and marked the wall with their inked middle fingertip. The difference between the two points was calculated as the final score.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali K, Gupta S, Hussain ME, Alzhrani M, Manzar MD, Khan M, Alghadir AH. Effect of plyometric versus complex training on core strength, lower limb, and upper limb power in male cricketers: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2023 Nov 27;15(1):160. doi: 10.1186/s13102-023-00771-8. PMID 38008712